CLINICAL TRIAL: NCT04544644
Title: A Phase II Study of AK104 (Binding Kenetics to PD-1 and CTLA-4) in Combination With Anlotinib in Patients With Advanced NSCLC
Brief Title: A Study of Combination Therapy in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weiwei Shi, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-001
Record Dates: First submitted 2020-08-29; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): AK104+anlotinib
  Interventions: Drug: AK104+anlotinib

INTERVENTIONS:
Drug: AK104+anlotinib — AK 104 is given by intravenous infusion and anlotinib is given by oral.

SUMMARY:
This trial is a single arm, two cohorts, phase II study. All patients are stage IIIB-IV NSCLC, Eastern Cooperative Oncology Group (ECOG) performance status 0-1 and no sensitizing mutation of the epidermal growth factor receptor gene or translocation of the anaplastic lymphoma kinase gene. Cohort 1 includes patients with metastatic or recurrent NSCLC after progression on treatment with platinum-based chemotherapy and PD-1/PD-L1, given concurrently or sequentially. Cohort 2 includes treatment naïve patients with advanced NSCLC. All patients will recieve AK104 15mg/kg every 3 weeks(for up to 2 years) and anlotinib(12mg/d). The primary end point are objective response rate per RECIST1.1 and safety. Secondary end points are progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years old (at the time consent is obtained);
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures);
* Have histologically- or cytologically-confirmed diagnosis of StageIIIB/C or IV NSCLC;
* Additional Inclusion Criteria for Cohort 1: Has metastatic or recurrent NSCLC after progression on treatment with platinum-based chemotherapy and PD-1/PD-L1, given concurrently or sequentially;
* Additional Exclusion Criteria for Cohort 2: Have no prior systemic chemotherapy for metastatic disease: at least 6 months since prior adjuvant chemotherapy;
* EGFR/ALK negative;
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy;
* Have a life expectancy of at least 3 months;
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team;
* Has adequate organ function as defined by: (1) Absolute neutrophil count >= 1,500/uL; (2) Platelets >= 100,000/uL; (3) Hemoglobin >= 9 g/dL; (4) Crcl >= 50ml/min; creatinine clearance may be calculated using the institutional/laboratory standard method; (5) Serum total bilirubin <= 1.5 ULN; (6) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 ULN; (7) Albumin >= 28g/L; (8) International Normalized Ratio (INR) and aPTT <1.5 ULN; (9) Left ventricular ejection fraction >= 50%;
* Have recovered from the effects of any prior radiotherapy or surgery;
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment;
* Has undergone major surgery within 30 days of Study Day 1;
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases;
* Has carcinomatous meningitis;
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
* Has an active infection requiring systemic therapy;
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study;
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy;
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment;
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  objective response rate per RECIST1.1

SECONDARY OUTCOMES:
PFS and OS | through study completion, an average of 2 years
  progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: weiwei Shi, Principal Investigator — Chinese PLA General Hospital